CLINICAL TRIAL: NCT02844127
Title: Effect of Right Ventricular Lead Position on Defibrillation Threshold
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices proposed for use in the protocol no longer used by physician
Sponsor: OhioHealth (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OhioHealth 16-0029
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apex First (Other): Patients born in odd-numbered years will receive an implantable cardioverter defibrillator (ICD). Defibrillation threshold determined with the right ventricular lead placed first in the apex and then in the septum. Final lead position will be determined at the discretion of the implanting physician.
  Interventions: Procedure: Implantable Cardioverter Defibrillator (ICD)
- Septum First (Other): Patients born in even-numbered years will receive an implantable cardioverter defibrillator (ICD). Defibrillation threshold determined with the right ventricular lead placed first in the septum and then in the apex. Final lead position will be determined at the discretion of the implanting physician
  Interventions: Procedure: Implantable Cardioverter Defibrillator (ICD)

INTERVENTIONS:
Procedure: Implantable Cardioverter Defibrillator (ICD) — Patients will receive an Implantable Cardioverter Defibrillator (ICD), with the leads implanted in either the apex or the septum as the first location. After defibrillation threshold is determined, the leads position will be changed to the second location and DFT will be determined again.

SUMMARY:
The purpose of this study is to determine how the position of the right ventricular (RV) coil of an implantable cardioverter defibrillator (apex versus septum) affects the defibrillation threshold; specifically, can defibrillator threshold be improved by implantation site selection.

DETAILED DESCRIPTION:
The investigators propose a prospective, pseudo-randomized study of patients who are electing to undergo implantation of an implantable cardioverter defibrillator (ICD).

There are two locations in the heart in which ICDs are normally implanted: the apex and the septum. The purpose of this study is to determine whether the ICD performs better in one location or the other, as measured by defibrillation threshold. In this study, both locations will be tested in each patient. The final location will be determined by the implanting physician as the location that is best for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicates for single-chamber (VR), dual-chamber (DR) or resynchronization CRT-D) implantable defibrillator
* Left-sided implant
* Single coil or dual coil (single coil for testing)
* Age ≥ 18 years of age
* Ability to consent
* Medically stable, in the opinion of the implanting physician, to undergo defibrillation safety margin testing
* Procedure performed under conscious sedation
* English-speaking

Exclusion Criteria:

* Patient unable to understand and consent to the procedure on his or her own
* Pregnant or breastfeeding patients
* New York Heart Association (NYHA) Class IV
* Patients with pre-existing RV leads
* Pacemaker dependent
* Patient medically unstable to undergo defibrillation testing (e.g., high risk for deep sedation; patients that develop respiratory compromise or hemodynamic instability from the sedation)
* Patients that require general anesthesia instead of conscious sedation
* Patients <18 years of age
* Non-English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Defibrillator threshold | At the time of each surgery through study completion, or up to 12 months
  Defibrillator threshold (DFT) will be determined at the time of implantation for each patient at the apex and the septum. A difference of >4 joules will be considered clinically significant.

SECONDARY OUTCOMES:
Percentage of patients with improved defibrillation threshold at the septum versus the apex | At the time of each surgery through study completion, or up to 12 months
  The percentage of patients that have an improved safety profile from septal implantation versus apical implantation will be calculated. Improved safety profile is defined as a defibrillation threshold increase of >4 joules.

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Rials, MD, PhD, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth Grant Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Because this is a pilot study with limited data collection, data will not need to be shared.